CLINICAL TRIAL: NCT07198009
Title: Modulation of Bioactive Lipids in Lipid Disorders: a Pilot Study of 2-HOBA Supplementation in Individuals With Elevated Lipoprotein(a)
Brief Title: 2-HOBA Supplementation in People With Elevated Lipoprotein(a)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2343236; 2343236 (Other Grant/Funding Number: Internal Grant)
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia; Elevated Lp(a)
Keywords: Oxidized Phospholipids; lp(a); 2HOBA
MeSH Terms: conditions — Hyperlipidemias | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-HOBA Supplementation for Elevated Lipoprotein(a) (Experimental): Participants will take oral 2-hydroxybenzylamine (2-HOBA, Hobamine) at a dose of 400 mg three times daily with meals for 6 weeks.
  Interventions: Dietary Supplement: 2-HOBA (Hobamine)

INTERVENTIONS:
Dietary Supplement: 2-HOBA (Hobamine) — Participants will take oral 2-hydroxybenzylamine (2-HOBA, Hobamine), a dietary supplement with Generally Recognized as Safe (GRAS) status. The study dose is 400 mg three times daily with meals for 6 weeks.

SUMMARY:
The goal of this clinical trial is to learn if a natural supplement called 2-hydroxybenzylamine (2-HOBA) can reduce harmful oxidized lipids and improve the function of lipoprotein(a) in adults with high lipoprotein(a) levels.

The main questions it aims to answer are:

Does 2-HOBA lower oxidized phospholipids on lipoprotein(a)? Does 2-HOBA reduce markers of inflammation and blood clotting in the blood?

Participants will:

Take 2-HOBA capsules (400 mg, three times daily with meals) for 6 weeks Provide blood and urine samples at the beginning, middle, and end of the study Have lab tests to measure changes in lipids, inflammation, and clotting markers

DETAILED DESCRIPTION:
Lipoprotein(a), or Lp(a), is a genetically determined cholesterol particle that increases the risk of heart disease and stroke. High levels of Lp(a) affect about 1 in 4 people, and there are no approved treatments that directly reduce its harmful effects. One reason Lp(a) is thought to be harmful is that it carries oxidized phospholipids, which promote inflammation and blood clotting.

2-hydroxybenzylamine (2-HOBA, also known as Hobamine) is a naturally occurring compound that neutralizes reactive molecules responsible for forming oxidized lipids. Preclinical studies and early human trials suggest that 2-HOBA is safe and may lower the buildup of oxidized phospholipids.

This pilot clinical trial will test whether oral 2-HOBA supplementation can improve the biology of Lp(a) in people with high levels (≥90 mg/dL). Ten adults will take 2-HOBA (400 mg by mouth, three times daily with meals) for 6 weeks. Blood and urine will be collected at three clinic visits (baseline, mid-study, and end of study). Researchers will measure oxidized phospholipids, lipoprotein function, markers of inflammation (such as C-reactive protein and interleukins), and markers of clotting (such as fibrinogen, D-dimer, and platelet activity).

The results will provide early information about whether 2-HOBA can reduce harmful changes linked to high Lp(a) and help guide the design of larger future trials.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-69 years.
* Elevated Lp(a) levels ≥ 90 mg/dL.
* Able to provide informed consent and adhere to study schedules.
* Willing to follow a physician-recommended diet during the study.

Exclusion Criteria:

* Pregnant, planning pregnancy during the study period, or currently breastfeeding.
* Individuals with established cardiovascular disease
* Planning major changes in diet or exercise routines.
* Experienced >20% weight change in the past 3 months.
* Diagnosed with malabsorption syndrome or chronic diarrhea.
* Abnormal liver, kidney, or thyroid function.
* Drug or alcohol abuse within the past 6 months, or significant mental/psychological impairment.
* Have known bleeding disorders (e.g., hemophilia).
* Planned surgery during the study period.
* Donated blood within the last 2 weeks or planning to donate during the study.
* Require regular blood transfusions.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in oxidized phospholipids (OxPL) on circulating lipoprotein(a) | 6 weeks
  OxPL levels on circulating lipoprotein(a) will be measured in blood samples collected before and after 6 weeks of oral 2-HOBA supplementation.

SECONDARY OUTCOMES:
High-sensitivity CRP | 6 weeks
  High-sensitivity CRP will be measured in blood samples to assess changes in systemic inflammation after 2-HOBA supplementation.
Interleukin-6 | 6 weeks
  IL-6 levels will be measured in plasma to evaluate the effect of 2-HOBA on inflammatory signaling.
Tumor Necrosis Factor-alpha (TNF-α) | 6 weeks
  TNF-α concentrations will be measured in plasma as an additional marker of inflammation.
Fibrinogen | 6 weeks
  Plasma fibrinogen levels will be measured to assess changes in blood clotting potential.
D-dimer | 6 weeks
  D-dimer will be measured in plasma as a marker of fibrinolysis and thrombosis.
Thromboxane | 6 weeks
  Urinary and plasma thromboxane B2 will be analyzed to evaluate platelet activation.
Platelet aggregation | 6 weeks
  Platelet aggregation will be measured using agonists such as arachidonic acid, ADP, and collagen.
Plasma Lp(a) concentrations | 6 weeks
  Plasma Lp(a) concentrations will be measured to monitor any effects of 2-HOBA on lipoprotein levels.

CONTACTS AND LOCATIONS:
Overall Officials: Wenliang Song, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- Lipid Clinic at Brown University Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No